CLINICAL TRIAL: NCT06402708
Title: Postoperative Adjuvant Treatment for Thymic Cancer With Completed Resection (Radiotherapy vs Chemoradiotherapy): A Prospective, Multicenter, Open-label, Phase III, Randomized Controlled Trial
Brief Title: Postoperative Adjuvant Chemotherapy for Thymic Cancer (FUSCC-Thymic 3)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kailiang Wu, professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2403293-1
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Thymic Carcinoma
Keywords: thymic carcinoma; adjuvant treatment; radiotherapy; chemotherapy
MeSH Terms: conditions — Thymoma | interventions — Drug Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy Arm (Active Comparator): Radiotherapy (50Gy/25f), IMRT
  Interventions: Radiation: Radiotherapy
- Chemoradiotherapy Arm (Experimental): 2 cycle of chemotherapy, and then radiotherapy of 50Gy/25f，and then another 2 cycle of chemotherapy
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — paclitaxel 60mg/m2, ivgtt; cisplatin 30mg/m2, ivgtt; 5-FU 500mg/m2, ivgtt and 500mg/m2, civ 24h; calcium folinate 200mg; q3w.
  Arms: Chemoradiotherapy Arm
Radiation: Radiotherapy — IMRT, 50Gy/25f
  Arms: Radiotherapy Arm

SUMMARY:
The goal of this clinical trial is to learn the role of adjuvant chemotherapy for patients with thymic carcinoma and completed resection. The main questions it aims to answer are:

1. Does adjuvant chemotherapy decrease disease progression?
2. Does medium dose of three drugs (paclitaxel, cisplatin, 5-FU) well tolerance?

Researchers will compare chemoradiotherapy to radiotherapy to see whether chemoradiotherapy could decrease disease progression or not.

Participants will:

1. Take radiotherapy (50Gy/25f) with or without 4 cycles of chemotherapy (TPF).
2. Follow up every 3 months in the first two year, and then every 6 months.

DETAILED DESCRIPTION:
Thymic carcinomas are rare neoplasms found in the anterior mediastinum, with an incidence of 0.38 cases per 100,000 people. Surgery is the primary treatment for patients with thymic carcinomas, and complete surgical resection proves fundamental for enhancing survival. However, the necessity for adjuvant therapy and the optimal type thereof for patients who have undergone complete resection remain unclear due to the lack of high-quality studies.

Our previous retrospective study found that radiotherapy improved overall survival and disease progression free survival significantly for all patients with thymic carcinoma and completed resection, however, chemotherapy only improved disease progression free survival for patients of stage III/IV. We also found that chemotherapy regimens containing paclitaxel were an advantageous combination for thymic cancer, and 1 or 2 cycles of adjuvant chemotherapy were better than more cycles, suggesting reduced dose chemotherapy.

DCF (docetaxel, cisplatin, 5-FU) or TPF (paclitaxel, cisplatin, 5-FU) were widely used in head and neck, esophageal, stomach, and anal canal cancer, and better effect were presented. However, the toxicity of full dose was too toxic to tolerate. Our previous experience in esophageal cancer found TPF with 2/3 of standard dose was well tolerance. Therefore, medium dose of TPF three drugs chemotherapy were chosed to balance efficacy and toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate and sign an informed consent form in writing;
2. Age range from 18 to 75 years old, regardless of gender;
3. Within 3 months after the surgery is completed;
4. Histologically diagnosed with thymic cancer;
5. Complete resection based on surgical records, pathological reports, and postoperative imaging;
6. Masaoka stage: I-III
7. No severe hematopoietic function, heart, lung, liver, kidney dysfunction, or immune deficiency;
8. White blood cells ≥ 3 × 109/L; Neutrophils ≥ 1.5 × 109/L; Hemoglobin ≥ 10 g/dL; Platelets ≥ 100 × 109/L; Total bilirubin ≤ 1.5 times the upper limit of normal value; AST (SGOT)/ALT (SGPT) ≤ 2.5 times the upper limit of normal value; Creatinine ≤ 1.5 times the upper limit of normal value;

Exclusion Criteria:

1. Having a second primary tumor (excluding cured non malignant melanoma of the skin, papillary thyroid carcinoma, stage I seminomatoma, cervical carcinoma in situ, or other curable tumors that have been tumor free for more than 3 years after treatment);
2. Symptomatic coronary heart disease, left heart failure, uncontrollable seizures, or loss of self-awareness due to mental illness;
3. Pregnancy and lactation period;
4. Patients with drug addiction, chronic alcoholism and AIDS;
5. Researchers believe that participants are not suitable for this experiment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 3 year
  From surgery to any disease relapse or death

SECONDARY OUTCOMES:
Overall survival | 3 year
  from surgery to any death
Disease Specific Survival | 3 year
  from surgery to death related to thymic carcinoma

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No